CLINICAL TRIAL: NCT03374540
Title: Comparative Effectiveness of Rivaroxaban and Warfarin for Stroke Prevention in Multi-morbid Patients With Nonvalvular Atrial Fibrillation
Brief Title: Rivaroxaban vs Warfarin for SPAF in Multi-morbid Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19859
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Nonvalvular Atrial Fibrillation
MeSH Terms: interventions — Rivaroxaban; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxaban: Patients who initiated Oral anticoagulant (OAC) treatment with rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Vitamin K antagonist (VKA): Patients who initiated OAC treatment with VKA
  Interventions: Drug: Vitamin K antagonist (VKA)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15/20 mg
  Groups: Rivaroxaban
Drug: Vitamin K antagonist (VKA) — Individually adjusted dose
  Groups: Vitamin K antagonist (VKA)

SUMMARY:
The overall goal of this study was to evaluate the comparative safety and effectiveness of rivaroxaban vs. vitamin K antagonist (VKA) for stroke prevention in patients with nonvalvular atrial fibrillation (NVAF) across risk profiles and comorbidities that reflect everyday clinical practice.

The primary objective in this study was to evaluate the combined end point of stroke or systemic embolism (SSE), and major bleeding in NVAF patients treated with rivaroxaban vs. VKA.

ELIGIBILITY:
Inclusion Criteria:

* Be oral anticoagulant naive during the 365 days before the day of the first qualifying oral anticoagulant (rivaroxaban or VKA) dispensing, and
* Have ≥365 days of continuous medical and prescription coverage before initiation of oral anticoagulation (which serves as the study's baseline period)

Exclusion Criteria:

* <18 years of age
* <2 International Classification of Diseases, Ninth/Tenth Revision, Clinical Modification diagnosis codes for atrial fibrillation
* Valvular heart disease
* Transient cause of NVAF
* Venous thromboembolism
* Hip or knee arthroplasty
* Malignant cancer
* Pregnancy
* >1 oral anticoagulant prescribed (on index date)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study will be all the insured individuals included in the Truven Health MarketScan Commercial Claims and Medicare Supplemental Databases (Truven MarketScan).
Sampling Method: Non-Probability Sample
Enrollment: 78517 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Stroke or systemic embolism (SSE) | Retrospective analysis from January 1, 2011 to December 31, 2017
Major bleeding | Retrospective analysis from January 1, 2011 to December 31, 2017
  Without access to clinical information and event adjudication in administrative claims data, major bleeding will operationalized as hospital-related bleeding using a clinically validated algorithm

SECONDARY OUTCOMES:
Hemorrhagic stroke | Retrospective analysis from January 1, 2011 to December 31, 2017
Ischemic stroke | Retrospective analysis from January 1, 2011 to December 31, 2017
Subtypes of major bleeding | Retrospective analysis from January 1, 2011 to December 31, 2017
Major adverse cardiovascular events (MACEs) and major adverse limb events (MALEs) | Retrospective analysis from January 1, 2011 to December 31, 2017
Acute kidney injury | Retrospective analysis from January 1, 2011 to December 31, 2017
Renal impairment | Retrospective analysis from January 1, 2011 to December 31, 2017

CONTACTS AND LOCATIONS:
Locations (1):
- Truven Health MarketScan Commercial Claims and Medicare Supplemental Databases, Multiple Locations, Washington, United States

REFERENCES:
- [Result] Coleman CI, Kreutz R, Sood N, Bunz TJ, Meinecke AK, Eriksson D, Baker WL. Rivaroxaban's Impact on Renal Decline in Patients With Nonvalvular Atrial Fibrillation: A US MarketScan Claims Database Analysis. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619868535. doi: 10.1177/1076029619868535. PMID 31392894
- [Result] Martinez BK, Baker WL, Sood NA, Bunz TJ, Meinecke AK, Eriksson D, Coleman CI. Influence of Polypharmacy on the Effectiveness and Safety of Rivaroxaban Versus Warfarin in Patients With Nonvalvular Atrial Fibrillation. Pharmacotherapy. 2019 Feb;39(2):196-203. doi: 10.1002/phar.2213. Epub 2019 Jan 28. PMID 30597611
- [Result] Baker WL, Beyer-Westendorf J, Bunz TJ, Eriksson D, Meinecke AK, Sood NA, Coleman CI. Effectiveness and safety of rivaroxaban and warfarin for prevention of major adverse cardiovascular or limb events in patients with non-valvular atrial fibrillation and type 2 diabetes. Diabetes Obes Metab. 2019 Sep;21(9):2107-2114. doi: 10.1111/dom.13787. Epub 2019 Jun 11. PMID 31099460
- [Result] Hernandez AV, Bradley G, Khan M, Fratoni A, Gasparini A, Roman YM, Bunz TJ, Eriksson D, Meinecke AK, Coleman CI. Rivaroxaban vs. warfarin and renal outcomes in non-valvular atrial fibrillation patients with diabetes. Eur Heart J Qual Care Clin Outcomes. 2020 Oct 1;6(4):301-307. doi: 10.1093/ehjqcco/qcz047. PMID 31432074